CLINICAL TRIAL: NCT00597441
Title: Phase I Study of Umbilical Cord Blood Transplantation Followed by Third Party Thymus Transplantation
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: accrual of evaluable subjects too low
Sponsor: Sumitomo Pharma Switzerland GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00007995
Record Dates: First submitted 2007-12-27; First posted 2008-01-18 (Estimated); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Stem Cell Transplantation
Keywords: unrelated; umbilical cord blood transplantation; thymus transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I (Experimental): Thymic tissue from third party donor
  Interventions: Biological: Thymic Transplantation for Recipients of UCB transplant

INTERVENTIONS:
Biological: Thymic Transplantation for Recipients of UCB transplant — Subjects with hematologic malignancies or bone marrow failure disorders will undergo umbilical cord blood transplantation and two months post transplant will have thymic tissue from a third party donor transplanted into the thigh muscle.

SUMMARY:
The objective of this trial is to assess the toxicity of thymus transplantation following unrelated umbilical cord blood transplantation. Emphasis will be placed on adverse events that are not typically associated with umbilical cord blood transplantation. Also, to determine whether engraftment of a third party thymus allograft is feasible in patients who have undergone unrelated umbilical cord blood transplantation.

DETAILED DESCRIPTION:
The objective of this trial is to assess the toxicity of thymus transplantation following unrelated umbilical cord blood transplantation. Emphasis will be placed on adverse events that are not typically associated with umbilical cord blood transplantation. Also, to determine whether engraftment of a third party thymus allograft is feasible in patients who have undergone unrelated umbilical cord blood transplantation. Thymic engraftment will be determined by biopsy of the thymus allograft and immunohistochemical evidence of thymopoiesis. In addition, we would like to assess thymic function by measuring the number of naive T cells and the number of T cell receptor rearrangement excision circles (TRECS), and by assessing the diversity of the T cell receptor beta chain. These data will be compared to age, stem-cell donor source and disease matched historical controls whose stem cell transplants were not followed by a thymus transplant. This will be done in descriptive fashion. Other immune parameters will be followed including T, B, and NK cell numbers, T cell responses to mitogens, antigens, and immunoglobulin production.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who received a dual cord blood transplant are eligible and must have achieved donor cord blood chimerism of > 75% in both T-cell and myeloid lineages
* At the time of thymus transplantation, subjects cannot have active grade II-IV acute graft versus host disease.
* At the time of thymus transplantation, the subject must have an absolute neutrophil count of > 500/ul and a platelet count of 50,000/ul (even if achieved via transfusion).
* At the time of thymus transplantation, the subject must have < or equal to 50 circulating CD 34+ cells/ul (as measured within 3 weeks of transplant date).
* At the time of thymus transplantation, subjects cannot be on greater than 2 mg/kg/day methylprednisolone or its equivalent of steroids.
* At the time of thymus transplantation, PT and PTT must be less that 1.5 times the ULN or must be correctable to this level.
* At the time of thymus transplantation, subjects cannot require oxygen or have pulmonary disease that would be thought to make general anesthesia a high risk.
* Subjects must be between the ages of 18 and 60 years of age.

Exclusion Criteria:

* Subjects cannot have bone marrow flow cytometry demonstrating residual leukemia
* Subjects cannot have insufficient subcutaneous tissue and muscle mass to be able to accept and heal a thymus transplant, as assessed by a surgeon.
* Prior to thymus transplantation, subjects cannot have evidence of active disease with HHV6, West Nile Virus, EBV, and CMV.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2005-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Toxicity of thymus transplantation following unrelated umbilical cord blood transplantation. Emphasis will be placed on adverse events that are not typically associated with umbilical cord blood transplantation. | 5 years

SECONDARY OUTCOMES:
To determine whether engraftment of a third party thymus allograft is feasible in patients who have undergone unrelated UCBT. Thymic engraftment will be determined by biopsy of the thymus allograft and immunohistochemical evidence of thymopoiesis. | 5 years
To assess thymic function by measuring the number of naive T cells and the number of T cell receptor rearrangement excision circles (TRECS), and by assessing the diversity of the T cell receptor beta chain. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Horwitz, MD, Principal Investigator — Duke Health; Mary L Markert, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States